CLINICAL TRIAL: NCT02748447
Title: Effects of Automated Adjustment of the Inspired Oxygen in Reducing the Risk of Regional Cerebral (rSO2) Hypo-oxygenation in Preterm Infants on Non Invasive or Invasive Respiratory Support
Brief Title: Automated Adjustment of Inspired Oxygen to Maintaining Regional Cerebral Oxygenation in Preterm Infants on Respiratory Support
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ASST Fatebenefratelli Sacco (Other)
Responsible Party: Principal Investigator, Gianluca Lista,MD, MD, ASST Fatebenefratelli Sacco
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PoloU
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Cerebrovascular Circulation; Premature Infants
MeSH Terms: conditions — Premature Birth

ARMS (2):
- A-FiO2 (Experimental): 24 hours in automated FiO2 adjustment to maintain SpO2 within a target range
  Interventions: Device: Automated FiO2 adjustment
- M-FiO2 (No Intervention): 24 hours in manual adjustment of FiO2 to maintain SpO2 within a target range

INTERVENTIONS:
Device: Automated FiO2 adjustment — AVEA ventilator according to SpO2 target range delivers an automated FiO2
  Arms: A-FiO2

SUMMARY:
Background: fluctuation of cerebral blood flow and oxygenation in neonates who undergo intensive care is an important risk factor for risk of neurodevelopmental impairment. Near infrared spectroscopy (NIRS) allow direct measurements of cerebral tissue oxygenation. Automated Fraction of Inspired Oxygen (FiO2) adjustment can maintain arterial oxygen saturation (SpO2) within a target range and may reduce risk of fluctuation of cerebral oxygenation.

Aim of this study: to evaluate the efficacy of automated FiO2 adjustment in maintaining SpO2 within a target range and in reducing the risk of cerebral tissue hypo-oxygenation due to SpO2 fluctuations in preterm infants on invasive or non invasive respiratory support with supplemental oxygen.

DETAILED DESCRIPTION:
Background: fluctuation of cerebral blood flow and oxygenation in neonates who undergo intensive care is an important risk factor for risk of neurodevelopmental impairment. Near infrared spectroscopy (NIRS) allow direct measurements of cerebral tissue oxygenation. Automated FiO2 adjustment can maintain arterial oxygen saturation (SpO2) within a target range and may reduce risk of fluctuation of cerebral oxygenation.

Aim of this study: to evaluate the efficacy of automated FiO2 adjustment in maintaining SpO2 within a target range and in reducing the risk of cerebral tissue hypo-oxygenation due to SpO2 fluctuations in preterm infants on invasive or non invasive respiratory support with supplemental oxygen.

Methodology: multicenter randomized cross-over clinical trial. The study will be carried out for almost 1 year .

Study centers: 7 Italian Neonatal Intensive Care Units (NICUs) Number of subjects: 60 infants to have a >90% power, with an alpha of p=0.01, of detecting a 5% difference in %-time in the target range and a 50% difference in both SpO2 hyperoxic and hypoxic %-time.

Diagnosis and main inclusion criteria: preterm infants of 25+0-28+6 weeks of gestational age, requiring invasive or non invasive respiratory support and supplemental oxygen.

Other enrollment requirements: All infants will be enrolled between >72 hours (end of transition period) and </= 7 days. Expected to remain of the current mode of support for the 48-hour intervention period. Infants with major congenital anomalies, haemodynamic instability (patent ductus arteriosus-PDA) or requiring catecholamines treatment, clinical evidence of seizures or ongoing sepsis (positive blood culture) during the study, or within 24 hours prior of enrollment, will be excluded.

Study product:AVEA ventilator with closed-loop inspired oxygen control (CLiO2) automated FiO2 control option. An additional sensor will be attached to the infant's forehead for continuous measurement of cerebral tissue oxygen saturation (rStO2) with 5100C NIRS oximeter, Covidien.

Duration:24 hours each of manual control and CLiO2 control. Reference therapy:Manual control of FiO2 provided according to standardized guidelines.

Statistical Methodology: repeated measures mixed linear model with control from sequence and ventilation mode.

Concurrent safety oversight:Independent Data Safety Monitoring Board, with blinded review every 6 months or 50% enrollment, and after 15 subjects.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants of 25+0-28+6 weeks of gestational age, requiring invasive or non invasive respiratory support and supplemental oxygen

Exclusion Criteria:

* infants with major congenital anomalies, haemodinamic instability, or requiring cathecolamines treatment,clinical evidence of seizures or ongoing sepsis (positive blood culture) during the study, or within 24 hours prior enrollment

Ages: 72 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-05 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
the burden of hypoxemia on regional cerebral saturation (rStO2) calculated as area under curve (AUC-% second) below the individual median rStO2 range ( defined as +/-5% of the individual rStO2 median of each infant during each period | 24 hours
  burden of hypoxemia on rStO2

SECONDARY OUTCOMES:
AUC above the individual median rStO2 and time (% of the total recording time) within the SpO2 target range (91-95%) | 24 hours
  burden hyperoxemia

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Lista, MD, Principal Investigator — ASST-FBF-Sacco
Locations (1):
- V. Buzzi Childrens's Hospital - ASST FBF-SACCO, Milan, Italy

REFERENCES:
- [Result] Kurth CD, McCann JC, Wu J, Miles L, Loepke AW. Cerebral oxygen saturation-time threshold for hypoxic-ischemic injury in piglets. Anesth Analg. 2009 Apr;108(4):1268-77. doi: 10.1213/ane.0b013e318196ac8e. PMID 19299799
- [Result] Laptook AR, Salhab W, Allen J, Saha S, Walsh M. Pulse oximetry in very low birth weight infants: can oxygen saturation be maintained in the desired range? J Perinatol. 2006 Jun;26(6):337-41. doi: 10.1038/sj.jp.7211500. PMID 16598294
- [Result] Claure N, D'Ugard C, Bancalari E. Automated adjustment of inspired oxygen in preterm infants with frequent fluctuations in oxygenation: a pilot clinical trial. J Pediatr. 2009 Nov;155(5):640-5.e1-2. doi: 10.1016/j.jpeds.2009.04.057. PMID 19595375
- [Result] van Kaam AH, Hummler HD, Wilinska M, Swietlinski J, Lal MK, te Pas AB, Lista G, Gupta S, Fajardo CA, Onland W, Waitz M, Warakomska M, Cavigioli F, Bancalari E, Claure N, Bachman TE. Automated versus Manual Oxygen Control with Different Saturation Targets and Modes of Respiratory Support in Preterm Infants. J Pediatr. 2015 Sep;167(3):545-50.e1-2. doi: 10.1016/j.jpeds.2015.06.012. Epub 2015 Jul 2. PMID 26144575